CLINICAL TRIAL: NCT04422600
Title: Fetal Exposure to Cannabinoids: Exposure, Methylation and Neurodevelopmental Effects
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 239611
Record Dates: First submitted 2020-05-28; First posted 2020-06-09 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2023-09

CONDITIONS: Fetal Exposure Timing Unspecified
Keywords: Fetal Exposure; Cannabinoids; Methylation; Neurodevelopmental Effects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Five (5) mL of blood will be collected from mothers at some point in the third trimester of pregnancy. Five (5) mL of umbilical cord blood will be collected from the baby immediately after birth, followed by a 1 mL venous blood sample collected 24 hours or later following birth during the routine blood sample collection for newborn screening.
  Buccal swabs will be collected from infants at 6 and 12 months of age for DNA methylation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Mothers who report use of THC with or without CBD: Mothers who report THC and CBD usage during the trimester month of pregnancy, at a frequency of at least three time per week. Information will be collected from mothers receiving their obstetrical care at UAMS and will include data on the exact products used and the frequency of use.
  Interventions: Other: There is no other intervention, only clinical treatment.
- Mothers who report use of CBD only: Mothers who report CBD usage during the trimester month of pregnancy, at a frequency of at least three time per week. Information will be collected from mothers receiving their obstetrical care at UAMS and will include data on the exact products used and the frequency of use.
  Interventions: Other: There is no other intervention, only clinical treatment.
- Control Mothers: Recruitment of pregnant women who do not use THC or CBD will be conducted using the Epic MyChart research participant recruitment tool
  Interventions: Other: There is no other intervention, only clinical treatment.

INTERVENTIONS:
Other: There is no other intervention, only clinical treatment. — The investigators will then correlate that exposure with neurodevelopmental outcomes.

SUMMARY:
Cannabis is a very popular drug for both recreational and medicinal use. An estimated 20% of adults in the United States report using cannabis in the past month, and this number continues to increase each year. As of 2018, medical use of cannabis is legal in 33 states and the District of Columbia. Recreational use is legal in 10 states, and it is decriminalized in 15 states. Hemp-derived cannabidiol (CBD) is legal in all states. Due to the rapidly changing legal status across the country, the demand for cannabinoids (which are specific components of cannabis), such as THC and CBD, are also rapidly increasing. Studies have shown a significant increase in marijuana use among pregnant and parenting women following state-wide legalization, and this could have significant implications for the health and development of children born to these women.

While there is a growing effort to evaluate the health effects of cannabinoids, especially during pregnancy, there is still relatively little known about the long term neurodevelopmental outcomes, such as emotional regulation, attention, and intelligence, in children born to mothers who used any sort of cannabinoid during pregnancy. The few studies that have been performed that look at longer term outcomes were epidemiological and self-reported in nature, and cannot accurately correlate neurodevelopmental outcomes with precise dosage and exposure levels during pregnancy.

Importantly, the THC content of marijuana has dramatically increased in recent years, with THC concentration and purity being the highest in history. It is estimated that cannabis potency has increased 3-fold over the past 2 decades. Many of the previous studies examining prenatal cannabis use and fetal outcomes reflected lower potency cannabis, which is not relevant to today's exposure levels. Additionally, there are no published studies to-date that evaluate fetal exposure to CBD or neurodevelopmental outcomes in infants who were exposed to CBD prenatally.

Finally, the causes behind possible neurodevelopmental changes in children exposed to cannabis prenatally have not been thoroughly explored, particularly in humans. It is thought that epigenetic modifications, or changes to DNA, may play a role in changes to the developing fetal brain after prenatal exposure to cannabis, but few studies have evaluated this quantitatively in humans.

DETAILED DESCRIPTION:
Cannabis is a very popular drug for both recreational and medicinal use. An estimated 20% of adults in the United States report using cannabis in the past month, and this number continues to increase each year. As of 2018, medicinal use of cannabis is legal in 33 states and the District of Columbia. Recreational use is legal in 10 states, and it is decriminalized in 15 states. Hemp-derived cannabidiol (CBD) is legal in all states. Due to the rapidly changing legal status across the country, the demand for tetrahydrocannabinoid (THC) and CBD products is also rapidly increasing. Studies have shown a significant increase in marijuana use among pregnant and parenting women following state-wide legalization, and this could have significant implications for the health and development of children born to these women.

Despite its widespread use, and increased interests in THC for medical treatment, significant gaps exist in the investigator's scientific knowledge of the pharmacology and pharmacokinetics of THC and its metabolites. When inhaled, THC and CBD reach maximum concentrations within seconds. Bioavailability varies widely and is a function of inhalation time, number, interval, and duration of puffs, as well as within product variability. Importantly, smokers have greater bioavailability of THC than non-smokers. When THC and CBD are orally consumed, the bioavailability is relatively low (< 20%). However, the lipophilicity of both THC and CBD make these compounds of great interest with respect to tissue distribution. CBD is more lipophilic than THC and thus more likely to be absorbed with topic application. THC is known to cross the placenta and can reach the fetus]. The metabolism of both THC and CBD is complex. Following absorption, THC and CBD are rapidly distributed to tissues with high blood flow. Metabolism occurs in the liver via CYP2C9, CYP2C19, and CYP3A4, as well as the brain, small intestine, heart and lung. Primary metabolites undergo glucuronidation or conjugation reactions. The elimination half-lives are prolonged due to the deposition of drug and metabolites in fat.

Some previous epidemiological studies have shown that children born to mothers who report using THC during their pregnancy have a higher prevalence of neurodevelopmental and behavioral abnormalities. While these studies are sparse, there have been some studies that follow longitudinal cohorts worldwide. These epidemiological, survey-based studies have reported an increase in executive functioning deficits in infants who were exposed to THC in utero. These studies have also shown an increase in attention problems and hyperactivity in these children during early childhood and later adolescence. However, these studies have reported inconsistent outcomes. Some have reported negative effects on cognitive or executive functioning, and others have reported no significant changes. One possibility for these discrepancies is that survey-based epidemiological studies do not accurately capture the exact levels of fetal exposure due to the unreliable nature of self-reporting, making it difficult to accurately correlate prenatal exposure levels to neurodevelopment. This makes the need for a well-designed, quantitative exposure study that is followed by longitudinal neurodevelopmental outcome measurement imperative to determining true correlations between prenatal THC use and developmental outcomes in children.

It has also previously been established that cannabis use during pregnancy can be detrimental to the developing fetus. Prenatal use of THC has been shown to cause low birth weight in the absence of any change in neonatal length or head circumference, as well as increased tremors and disrupted sleep patterns. It has also been correlated with an increased need for placement in the neonatal intensive care unit. In addition to human studies, animal studies have shown changes in the endocannabinoid system (ECS) in the fetal brain during development. The ECS is present in the developing brain from the time of 5 weeks gestation, and is required for proliferation, differentiation, and migration of neurons. Any changes to this system during development could have important implications for further neural development. Several studies have observed changes in postsynaptic target selectivity, differentiation of developing axons, and disruption of position in the ECS in animal fetuses that were exposed to THC in utero. These central nervous system alterations could potentially point to long-term neurodevelopmental changes in children born to mothers who used cannabis during pregnancy. However, while animal studies are able to report exact dosing levels, animal models of prenatal cannabinoid use often do not accurately reflect human use.

While some detrimental effects to the fetus following prenatal cannabis use have been observed in both animal models and human studies, there remains the mechanistic question of what is causing these changes. Some studies have proposed epigenetic reprogramming that may occur in the mothers and the babies following prenatal cannabis use. Prior studies have focused on the effects of prenatal cannabis use increasing the likelihood of the children's substance abuse later in life, and have found positive correlations to DNA methylation and histone modification in these cases. Additionally, it has been shown that paternal cannabis use alters DNA methylation in sperm of rats and humans, which could also have important implications for development. However, to-date, there have not been any studies correlating epigenetic changes and neurodevelopmental changes in infants prenatally exposed to cannabis.

Additionally, many of the prior human studies were done at a time when THC content in marijuana was not as high as is in today's market, which could have major implications for actual exposure levels in the fetus. The initial studies that evaluated the effects of prenatal cannabis use on fetal outcomes were done in the early 1990s, at a time when average THC potency in seized marijuana in the United States was approximately 4%. The most recently reported potency of seized illicit cannabis plant material is approximately 12%. Additionally, the ratio of psychoactive THC content to non-psychoactive cannabidiol content has increased from approximately 14 to 80 between 1995 and 2014. These factors suggest a need for more updated studies that examine the effects of current high potency levels of fetal exposure to cannabis, as an increase in potency may have greater effects on the developing fetus.

While there have been some prior studies measuring the effects of fetal exposure to THC specifically, there have been no studies to-date that have evaluated the effects of CBD exposure on the developing fetus. CBD (also known as hemp) supposedly lacks psychoactive THC components, making it legal, widely available, and generally perceived to be safe.CBD is touted as a treatment for a number of conditions, including depression, anxiety, pain, and cancer. These factors, in addition to strong marketing campaigns, have most likely caused an increase in prenatal CBD use in recent years. A recent study conducted in mice found that CBD activates a large range of CYPP450 enzymes. While these data are preliminary, CYPP450 activation raises the concern of drug-drug interactions and suggests that biologic activity of CBD is not fully understood. However, there are no published studies evaluating the effects of prenatal CBD use on fetal outcomes or neurodevelopment. Additionally, many CBD products have been shown to contain varying concentrations of CBD, or are contaminated with synthetic cannabinoids (e.g. K2, "spice") or THC. The investigators will establish the exact composition of the products the pregnant women are taking in order to properly evaluate potential exposure levels in the developing fetus. The investigators will then correlate that exposure with neurodevelopmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Age 18 and older
* Must plan to give birth at UAMS
* Report regular (at least 3x per week) use of THC- and/or CBD-containing product anytime during pregnancy (for experimental groups). Women who discontinue use of marijuana and/or CBD during pregnancy will still be allowed in the study.
* Pregnant women who do not use THC or CBD will be enrolled as controls.

Exclusion Criteria:

* Any other illicit drug use during pregnancy
* Plan to give birth anywhere other than UAMS

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women and infants
Study Population: Mothers who report use of THC and /or CBD and pregnant women who do not use THC or CBD. Babies will be enrolled (consent given by mothers) following birth.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
THC and CBD metabolite levels in maternal neonatal blood | Within three months prior to the estimated due date
  Levels of THC and CBD metabolites will be measured in maternal blood following prenatal drug use. These levels will be measured via liquid chromatography-mass spectrometry.
THC and CBD metabolite level in umbilical cord blood | Immediately after birth
  Levels of THC and CBD metabolites will be measured umbilical cord blood following prenatal drug use. These levels will be measured via liquid chromatography-mass spectrometry.
THC and CBD metabolite levels in neonatal blood | 24 hours after birth
  Levels of THC and CBD metabolites will be measured in neonatal blood following prenatal drug use. These levels will be measured via liquid chromatography-mass spectrometry.
Infant motor, cognitive, and social development at 6 months of age using the Ages and Stages Questionnaire | 6 months after birth
  To measure infant neurodevelopment, we will use the Ages and Stages Questionnaire (ASQ). The ASQ measures 5 domains/scales of child development: communication, gross motor, fine motor, problem solving, and personal-social. Each scale ranges from 0 to 60, with lower scores being indicative of deficits or poor outcomes.
Infant motor, cognitive, and social development at 12 months of age using the Ages and Stages Questionnaire | 12 months after birth
  To measure infant neurodevelopment, we will use the Ages and Stages Questionnaire (ASQ). The ASQ measures 5 domains/scales of child development: communication, gross motor, fine motor, problem solving, and personal-social. Each scale ranges from 0 to 60, with lower scores being indicative of deficits or poor outcomes.
Infant motor, cognitive, and social development at 6 months of age using the Bayley Scales of Infant Development | 6 months after birth
  To measure infant neurodevelopment, we will use the Bayley Scales of Infant and Toddler Development. The Bayley Scales measures 5 domains of child development: adaptive behavior, cognitive, language, motor, and social-emotional. Each scale ranges from 40-160, with higher scores indicative of better outcomes.
Infant motor, cognitive, and social development at 12 months of age using the Bayley Scales of Infant Development | 12 months after birth
  To measure infant neurodevelopment, we will use the Bayley Scales of Infant and Toddler Development. The Bayley Scales measures 5 domains of child development: adaptive behavior, cognitive, language, motor, and social-emotional. Each scale ranges from 40-160, with higher scores indicative of better outcomes.
DNA methylation profiles in infants at 12 months of age | 12 months after birth
  Buccal samples from infants at 12 months of age will be used to evaluate DNA methylation profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Kennon McGill, Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Hasin DS. US Epidemiology of Cannabis Use and Associated Problems. Neuropsychopharmacology. 2018 Jan;43(1):195-212. doi: 10.1038/npp.2017.198. Epub 2017 Aug 30. PMID 28853439
- [Background] Grant TM, Graham JC, Carlini BH, Ernst CC, Brown NN. Use of Marijuana and Other Substances Among Pregnant and Parenting Women With Substance Use Disorders: Changes in Washington State After Marijuana Legalization. J Stud Alcohol Drugs. 2018 Jan;79(1):88-95. PMID 29227236
- [Background] Goncalves J, Rosado T, Soares S, Simao AY, Caramelo D, Luis A, Fernandez N, Barroso M, Gallardo E, Duarte AP. Cannabis and Its Secondary Metabolites: Their Use as Therapeutic Drugs, Toxicological Aspects, and Analytical Determination. Medicines (Basel). 2019 Feb 23;6(1):31. doi: 10.3390/medicines6010031. PMID 30813390
- [Background] Grotenhermen F. Pharmacokinetics and pharmacodynamics of cannabinoids. Clin Pharmacokinet. 2003;42(4):327-60. doi: 10.2165/00003088-200342040-00003. PMID 12648025
- [Background] McLemore GL, Richardson KA. Data from three prospective longitudinal human cohorts of prenatal marijuana exposure and offspring outcomes from the fetal period through young adulthood. Data Brief. 2016 Oct 18;9:753-757. doi: 10.1016/j.dib.2016.10.005. eCollection 2016 Dec. PMID 27833935
- [Background] Calvigioni D, Hurd YL, Harkany T, Keimpema E. Neuronal substrates and functional consequences of prenatal cannabis exposure. Eur Child Adolesc Psychiatry. 2014 Oct;23(10):931-41. doi: 10.1007/s00787-014-0550-y. Epub 2014 May 3. PMID 24793873
- [Background] Day NL, Leech SL, Goldschmidt L. The effects of prenatal marijuana exposure on delinquent behaviors are mediated by measures of neurocognitive functioning. Neurotoxicol Teratol. 2011 Jan-Feb;33(1):129-36. doi: 10.1016/j.ntt.2010.07.006. PMID 21256427
- [Background] Fried PA. The Ottawa Prenatal Prospective Study (OPPS): methodological issues and findings--it's easy to throw the baby out with the bath water. Life Sci. 1995;56(23-24):2159-68. doi: 10.1016/0024-3205(95)00203-i. PMID 7539879
- [Background] Warshak CR, Regan J, Moore B, Magner K, Kritzer S, Van Hook J. Association between marijuana use and adverse obstetrical and neonatal outcomes. J Perinatol. 2015 Dec;35(12):991-5. doi: 10.1038/jp.2015.120. Epub 2015 Sep 24. PMID 26401751
- [Background] Gunn JK, Rosales CB, Center KE, Nunez A, Gibson SJ, Christ C, Ehiri JE. Prenatal exposure to cannabis and maternal and child health outcomes: a systematic review and meta-analysis. BMJ Open. 2016 Apr 5;6(4):e009986. doi: 10.1136/bmjopen-2015-009986. PMID 27048634
- [Background] Ko JY, Tong VT, Bombard JM, Hayes DK, Davy J, Perham-Hester KA. Marijuana use during and after pregnancy and association of prenatal use on birth outcomes: A population-based study. Drug Alcohol Depend. 2018 Jun 1;187:72-78. doi: 10.1016/j.drugalcdep.2018.02.017. Epub 2018 Mar 29. PMID 29627409
- [Background] Huizink AC. Prenatal cannabis exposure and infant outcomes: overview of studies. Prog Neuropsychopharmacol Biol Psychiatry. 2014 Jul 3;52:45-52. doi: 10.1016/j.pnpbp.2013.09.014. Epub 2013 Sep 27. PMID 24075896
- [Background] Metz TD, Allshouse AA, Hogue CJ, Goldenberg RL, Dudley DJ, Varner MW, Conway DL, Saade GR, Silver RM. Maternal marijuana use, adverse pregnancy outcomes, and neonatal morbidity. Am J Obstet Gynecol. 2017 Oct;217(4):478.e1-478.e8. doi: 10.1016/j.ajog.2017.05.050. Epub 2017 May 31. PMID 28578174
- [Background] Feldman RM. Smokeless tobacco spoils more than the world series. Todays FDA. 1990 Dec;2(12):1D. No abstract available. PMID 2288786
- [Background] Vargish GA, Pelkey KA, Yuan X, Chittajallu R, Collins D, Fang C, McBain CJ. Persistent inhibitory circuit defects and disrupted social behaviour following in utero exogenous cannabinoid exposure. Mol Psychiatry. 2017 Jan;22(1):56-67. doi: 10.1038/mp.2016.17. Epub 2016 Mar 15. PMID 26976041
- [Background] de Salas-Quiroga A, Diaz-Alonso J, Garcia-Rincon D, Remmers F, Vega D, Gomez-Canas M, Lutz B, Guzman M, Galve-Roperh I. Prenatal exposure to cannabinoids evokes long-lasting functional alterations by targeting CB1 receptors on developing cortical neurons. Proc Natl Acad Sci U S A. 2015 Nov 3;112(44):13693-8. doi: 10.1073/pnas.1514962112. Epub 2015 Oct 12. PMID 26460022
- [Background] Trezza V, Cuomo V, Vanderschuren LJ. Cannabis and the developing brain: insights from behavior. Eur J Pharmacol. 2008 May 13;585(2-3):441-52. doi: 10.1016/j.ejphar.2008.01.058. Epub 2008 Mar 18. PMID 18413273
- [Background] Szutorisz H, Hurd YL. High times for cannabis: Epigenetic imprint and its legacy on brain and behavior. Neurosci Biobehav Rev. 2018 Feb;85:93-101. doi: 10.1016/j.neubiorev.2017.05.011. Epub 2017 May 12. PMID 28506926
- [Background] Cecil CA, Walton E, Smith RG, Viding E, McCrory EJ, Relton CL, Suderman M, Pingault JB, McArdle W, Gaunt TR, Mill J, Barker ED. DNA methylation and substance-use risk: a prospective, genome-wide study spanning gestation to adolescence. Transl Psychiatry. 2016 Dec 6;6(12):e976. doi: 10.1038/tp.2016.247. PMID 27922636
- [Background] DiNieri JA, Wang X, Szutorisz H, Spano SM, Kaur J, Casaccia P, Dow-Edwards D, Hurd YL. Maternal cannabis use alters ventral striatal dopamine D2 gene regulation in the offspring. Biol Psychiatry. 2011 Oct 15;70(8):763-769. doi: 10.1016/j.biopsych.2011.06.027. Epub 2011 Aug 5. PMID 21820648
- [Background] Murphy SK, Itchon-Ramos N, Visco Z, Huang Z, Grenier C, Schrott R, Acharya K, Boudreau MH, Price TM, Raburn DJ, Corcoran DL, Lucas JE, Mitchell JT, McClernon FJ, Cauley M, Hall BJ, Levin ED, Kollins SH. Cannabinoid exposure and altered DNA methylation in rat and human sperm. Epigenetics. 2018;13(12):1208-1221. doi: 10.1080/15592294.2018.1554521. Epub 2018 Dec 18. PMID 30521419